CLINICAL TRIAL: NCT01153581
Title: Sex Hormones and Orthostatic Tolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0512000875a; 2R01HL071159-04 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Orthostatic Intolerance
MeSH Terms: conditions — Orthostatic Intolerance | interventions — ganirelix; Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ganirelix acetate (Experimental): Subjects were given 250 μg in 0.5ml normal saline for 16 days. (Organon, Roseland, NJ, USA)
  Interventions: Drug: Ganirelix acetate
- 17β-Oestradiol, E2 (Experimental): The same women added 17β-Oestradiol, E2; 0.2 mg day-1 patch (Vivelle; CIBA Pharmaceuticals, Summit, NJ) for days 4-16.
  Interventions: Drug: 17β-Oestradiol
- Progesterone (Experimental): The same women added progesterone (P4, 200 mg day-1 Prometrium, oral, Solvay Pharmaceuticals, Marietta, GA, USA) on days 13-16.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Ganirelix acetate — Ganirelix acetate: .25 ml/day by subcutaneous injection
  Other Names: Antagon
  Arms: Ganirelix acetate
Drug: 17β-Oestradiol — 17 beta estradiol: 0.2 mg/day (patches)
  Other Names: 17 beta estradiol; estradiol
  Arms: 17β-Oestradiol, E2
Drug: Progesterone — progesterone, 200 mg day-1 oral
  Other Names: P4; Prometrium
  Arms: Progesterone

SUMMARY:
This study is designed to determine the causes of "orthostatic intolerance" which occurs more commonly in women than in men. Orthostatic tolerance is the ability to remain standing up right for long periods of time, or to avoid dizziness when moving to standing from a seated or lying position.

DETAILED DESCRIPTION:
In this study we are interested in determining the impact of female reproductive hormones (estrogen and progesterone) on orthostatic tolerance (described above) so we administer these hormones to participants. We also test participants' orthostatic tolerance in our laboratory and use this information to place subjects into groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, English-speaking non-smoking women age 18- 34 with regular menses

Exclusion Criteria:

* Gynecologic:

  1. current or past estrogen-dependent neoplasia,
  2. unexplained vaginal bleeding,
  3. history of uterine fibroids,
  4. current pregnancy,
  5. known or suspected breast or uterine cancer,
  6. partial or complete hysterectomy
* Cardiac:

  1. myocardial infarction, ventricle tachycardia or fibrillation,
  2. angina,
  3. valvular disease,
  4. congestive heart failure, orthopnea, paroxysmal nocturnal dyspnea,
  5. current arrhythmias,
  6. prosthetic valves
* Pulmonary:

  1. current cigarette smokers, or pipe or cigar smokers,
  2. chronic obstructive pulmonary disease,
  3. adult asthma,
  4. dyspnea on exertion,
  5. current bronchitis, pneumonia, or tuberculosis,
  6. lung carcinoma,
  7. pulmonary embolus, recent
* Vascular:

  1. claudication or history of peripheral vascular disease,
  2. abdominal or thoracic aortic aneurysm, or repair of same,
  3. cerebral aneurysm, vascular malformations,
  4. hypertension, systolic or diastolic, or strong family history of hypertension
* Gastrointestinal:

  1. GI malignancy,
  2. hepatitis, current,
  3. splenomegaly from any cause,
  4. Cholecystitis,
  5. current diverticulosis or diverticulitis, inflammatory bowel disease, ulcerative colitis, Crohn's Disease,
  6. previous gastrointestinal surgery
* Infectious Disease: any intercurrent infection
* Hematologic/Oncologic:

  1. receiving chemotherapy or radiation therapy,
  2. any metastatic malignancy,
  3. anemia (hematocrit < 35),
  4. thrombocytopenia or thrombocytosis,
  5. neutropenia,
  6. hematologic malignancy,
  7. bleeding dyscrasia
* Neurologic:

  1. history of cerebral vascular accident with any neurologic sequels,
  2. uncontrolled seizures (e.g. more than 1 seizure/year),
  3. transient ischemic attacks,
  4. dementia,
  5. neurologic conditions producing dyscoordination, peripheral neuropathy, or myopathy,
  6. severe migraine headaches
* Endocrine:

  1. diabetes mellitus,
  2. any untreated endocrinopathy
* Renal:

  1. chronic renal disease,
  2. any history of renal disease or impairment,
  3. current urinary tract infection
* Musculoskeletal:

  1. inflammatory arthritis history (e.g., rheumatoid, psoriatic, Reiters),
  2. any history of pathologic fractures, including vertebral compression fractures
* Pharmacologic:

  1. any illegal drug use,
  2. alcohol use greater than an average of 4 oz/day over 30 days,
  3. coumadin or heparin use,
  4. current systemic antifungal use

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2006-02; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Stachenfeld, PhD, Principal Investigator — Yale University
Locations (1):
- John B. Pierce Laboratory, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
Our data are stored in locked files, and our spreadsheets and raw data are available should they be requested

RESULTS

PARTICIPANT FLOW:
Groups:
- Women With and Without Orthostatic Intolerance: Estrogen and Progesterone
  17 beta estradiol, progesterone, ganirelix acetate: Antagon (for ganirelix acetate)--0.25 ml per day, subcutaneous injection estradiol 0.2 mg/day (patches) per day progesterone 200 mg per day, pills
  17 beta estradiol, progesterone, ganirelix acetate: 17 beta estradiol: 0.2 mg/day (patches) progesterone 200 mg/day ganirelix acetate 0.25 mg/day
Period: Overall Study
Arm/Group | Women With and Without Orthostatic Intolerance
Started | 109
Completed | 109
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Women: Estrogen and Progesterone
  17 beta estradiol, progesterone, ganirelix acetate: Antagon (for ganirelix acetate)--0.25 ml per day, subcutaneous injection estradiol 0.2 mg/day (patches) per day progesterone 200 mg per day, pills
  17 beta estradiol, progesterone, ganirelix acetate: 17 beta estradiol: 0.2 mg/day (patches) progesterone 200 mg/day ganirelix acetate 0.25 mg/day
Arm/Group | Women
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 109
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 48
  More than one race | 3
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Orthostatic Tolerance
Description: We used a measure called cumulative stress index to determine orthostatic tolerance, which is the amount of time at a level of negative pressure each subject can maintain before feeling as if she is going to pass out. This is calculated by multiplying the pressure in mm Hg by the time in min.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: mmHg*min
Arm/Group | Women With and Without Orthostatic Intolerance
Number analyzed (Participants) | 109
mmHg*min | 634 (213)

2. Primary Outcome: Baroreceptor Function
Description: This is a measure of how the body responds to changes in pressure induced by changes in position such as sitting, lying standing. The pressure changes are induced by gravity. The measurement described below to assess baroreceptor function is units of change in forearm vascular resistance for a given change in lower body negative pressure. This allows us to determine how good the body is at sending signals to the periphery to respond to postural changes.
  Baroreflex sensitivity is defined as the change in interbeat interval (IBI) in milliseconds per unit change in BP. For example, when the BP rises by 10 mmHg and IBI increases by 100 ms, BRS would be 100/10 = 10 ms/mmHg.
Time Frame: 2 months
Population: Women with low and high orthostatic tolerance
Measure: Mean (Standard Error); unit: ms/mm Hg
Groups:
- Low Orthostatic Tolerance: Women who pass out easily in response to posture change
- High Orthostatic Tolerant: Women who can tolerate posture changes
Arm/Group | Low Orthostatic Tolerance | High Orthostatic Tolerant
Number analyzed (Participants) | 7 | 7
ms/mm Hg | 0.140 (0.034) | 0.128 (0.044)

3. Primary Outcome: Skin Microvascular Responses
Description: Changes in blood flow in the small vessel in the skin are measured in response to sequential heat and drug stimulation. It is measured in volts, and then corrected for a maximum level and expressed as "% max." This is measured with a Laser Doppler probes, which measures volts.
Time Frame: 2 months
Population: Women with and without orthostatic intolerance
Measure: Mean (Standard Error); unit: Percent of max volts
Groups:
- Women With Orthostatic Intolerance: Estrogen and Progesterone
  17 beta estradiol, progesterone, ganirelix acetate: Antagon (for ganirelix acetate)--0.25 ml per day, subcutaneous injection estradiol 0.2 mg/day (patches) per day progesterone 200 mg per day, pills
  17 beta estradiol, progesterone, ganirelix acetate: 17 beta estradiol: 0.2 mg/day (patches) progesterone 200 mg/day ganirelix acetate 0.25 mg/day
- Women Without Orthostatic Tolerance: Women who pass out easily with gravitational challenge
Arm/Group | Women With Orthostatic Intolerance | Women Without Orthostatic Tolerance
Number analyzed (Participants) | 8 | 8
Percent of max volts | 4.02 (0.39) | 5.18 (0.31)
Statistical Analysis 1: Comparison: Women With Orthostatic Intolerance vs Women Without Orthostatic Tolerance; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = -1.16

ADVERSE EVENTS:
Time Frame: 4 years
Groups:
- Ganirelix Acetate: Ganirelix acetate (Organon, Roseland, NJ, USA), a synthetic decapeptide with high antagonistic activity against naturally occurring gonadotrophin-releasing hormone (GnRH) to suppress GnRH. (250 μg in 0.5ml normal saline for 16 days).
- 17β-Oestradiol: The same women added 17β-Oestradiol, E2; 0.2 mg day-1 patch (Vivelle; CIBA Pharmaceuticals, Summit, NJ) for days 4-16.
Arm/Group | Ganirelix Acetate | 17β-Oestradiol | Progesterone
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/109 | 0/109
Other Adverse Events (participants affected / at risk) | 0/109 | 0/109 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other